CLINICAL TRIAL: NCT01711697
Title: An Alternative Radiation Fractionation Strategy for Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Emory University (Other)
Collaborators: Washington University Siteman Cancer Center (Other)
Responsible Party: Principal Investigator, Kristin Higgins, MD, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00056552; NCI-2012-01934 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD2179-12 (Other: Winship Cancer Institute)
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Carboplatin; Paclitaxel; Taxes; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiation therapy, carboplatin, paclitaxel, SBRT) (Experimental): Patients undergo radiation therapy daily and receive carboplatin and paclitaxel weekly for 4.5 weeks. Patients then undergo 2 boost SBRT treatments 2-3 days apart.
  Interventions: Radiation: stereotactic body radiation therapy; Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
Drug: carboplatin
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: paclitaxel
  Other Names: Anzatax; Asotax; TAX; Taxol
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
This phase I trial studies the best dose of radiation therapy in treating patients with locally advanced non-small cell lung cancer that cannot be removed by surgery. Radiation therapy uses high energy x rays to kill tumor cells. Specialized radiation therapy, such as stereotactic body radiation therapy (SBRT), that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. SBRT has been shown to provide excellent results when used in early stage lung cancer, but has not yet been applied to patients with more advanced disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To test the safety and tolerability of an alternative fractionation regimen in locally advanced non-small cell lung cancer (NSCLC), consisting of 44 Gy with concurrent chemotherapy followed by a stereotactic body radiation therapy (SBRT) boost to remaining parenchymal and nodal disease. The maximum tolerated dose of the SBRT boost will be determined.

SECONDARY OBJECTIVES:

1. To assess local control.
2. To assess distant metastasis and patterns of failure.
3. To assess overall survival at 1 and 2 years.

OUTLINE: This is a dose-escalation study of radiation therapy and SBRT.

Patients undergo radiation therapy daily and receive carboplatin and paclitaxel weekly for 4.5 weeks. Patients then undergo 2 boost SBRT treatments 2-3 days apart.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven NSCLC, within 8 weeks prior to patient registration
* Unresectable disease
* Clinical stage Tx, T1-T4, N1-3, M0
* Karnofsky performance status (KPS) ≥ 70
* Pretreatment positron emission tomography (PET) CT scan to rule out metastatic disease

  * The primary tumor may not be larger than 8 cm in maximum dimension
  * If the primary tumor is central in location, defined as within 2 cm from the tracheobronchial tree, it must be no larger than 5 cm
  * Mediastinal and hilar lymphadenopathy can be no larger than 5 cm at any nodal station
* Pretreatment brain CT with contrast or brain MRI to rule out metastases
* Pathologic assessment of the mediastinum to document involved nodal stations
* All of the above inclusion criteria must occur within 8 weeks prior to patient registration, with the exception of pathologic assessment of the mediastinum and biopsy to confirm NSCLC, which can be done within 12 weeks of patient registration

Exclusion Criteria:

* Prior history of lung cancer
* Pregnancy
* Prior history of radiation to the chest

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09-04 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) defined to be the dose level that results in a probability equal to 0.33 that a dose limiting toxicity (DLT) will be manifest using Common Terminology Criteria for Adverse Events (CTCAE) version 4 (v.4) | Up to 1 year
Acute toxicities associated with this regimen using CTCAE v.4 | Up to 90 days
  Crude rates of grade 3 and greater acute toxicities will be reported.
Late toxicities associated with this regimen using CTCAE v.4 | After 90 days
  Crude rates of grade 3 and greater late toxicities will be reported.

SECONDARY OUTCOMES:
Local control | Up to 5 years
  Will be calculated for the entire cohort using Kaplan-Meier methodology.
Distant metastasis | Up to 5 years
  Will be calculated for the entire cohort using Kaplan-Meier methodology.
Patterns of failure | Up to 5 years
  Will be assessed with standard follow-up imaging, and the percentages of in-field failures versus regional nodal failures calculated.
Overall survival | At 1 year
  Will be calculated for the entire cohort using Kaplan-Meier methodology.
Overall survival | At 2 years
  Will be calculated for the entire cohort using Kaplan-Meier methodology.
Overall survival | At 5 years
  Will be calculated for the entire cohort using Kaplan-Meier methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Higgins, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Siteman Cancer Center - Washington University, St Louis, Missouri